CLINICAL TRIAL: NCT03405181
Title: Effects of the Additional Weight on the Reaching Behavior of Preterm Infants With Low Birth Weight: Randomized Controlled Trial
Brief Title: Effects of the Additional Weight on the Reaching Behavior of Pre Term Infants With Low Birth Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Prof. Rodrigo Luiz Carregaro, Prof. Dr., University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Additional Weight Trial
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Preterm Infant; Infant Development; Low Birth Weight
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor won't have any knowledge about the study purposes and will be unaware of the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training with additional weight (Experimental): The infants will be submitted to a reaching behavior training program of 4 weeks, two times per week (totaling 8 sessions). During this training program, infants will use a bracelet with an additional weight characterized by 20% of the total mass of the upper limb placed on both wrists. This training will be adopted for the adequate weight intervention group and low weight intervention group.
  Interventions: Other: Training with additional weight
- Training without additional weight (Placebo Comparator): The infants will be submitted to a reaching behavior training program of 4 weeks, two times per week (totaling 8 sessions). During this training program, infants will use a bracelet without additional weight, placed on both wrists. This training will be adopted for the adequate weight placebo group and low weight placebo group.
  Interventions: Other: Training without additional weight

INTERVENTIONS:
Other: Training with additional weight — The infants will be positioned in a reclined position. A bracelet with an additional weight (20% of the total mass of the upper limb) will be placed on both wrists. The training will happen 2x/week, during 4 weeks (8 sessions). An object will be used to stimulate the reaching behavior, which will be displayed by the examiner (positioned in front of the infant), and presented in the midline at shoulder height, considering the distance from the arm's length of the infant to the height of the wrist. The physiotherapist will draw the attention of the infant to the object, moving it momentarily so that the infant perceives it and reaches it. After reaching, the object will be carefully removed and resubmitted in order to elicit a new movement. The interval between each presentation will be of approximately 5 seconds. At least 10 movements will be stimulated. If the infant does not achieve the 10 reaches within the maximum interval of 15 minutes, the session will be terminated.
  Arms: Training with additional weight
Other: Training without additional weight — The infants will be positioned in a reclined position. A bracelet without the additional weight will be placed on both wrists. The training will happen 2x/week, during 4 weeks (8 sessions). An object will be used to stimulate the reaching behavior, which will be displayed by the examiner (positioned in front of the infant), and presented in the midline at shoulder height, considering the distance from the arm's length of the infant to the height of the wrist. The physiotherapist will draw the attention of the infant to the object, moving it momentarily so that the infant perceives it and reaches the object. After reaching, the object will be carefully removed (or picked up) and resubmitted in order to elicit a new movement. The interval between each presentation of the object will be of approximately 5 seconds. At least 10 movements will be stimulated. If the infant does not achieve the 10 reaches within the maximum interval of 15 minutes, the session will be terminated.
  Arms: Training without additional weight

SUMMARY:
The effects of additional weight on early motor skills of infants have been increasingly studied. During the reaching behavior, the additional weight has been shown benefits in certain kinematic variables in full term and preterm infants. There is a growing interest in the study of populations at risk for motor development, especially considering interventions based on functional activities with the purpose of improving the neuromotor control, functional capacity and muscle strength. The aim of the present study is to investigate the effect of a functional training with additional weight in the reaching behavior of preterm infants with low birth weight and to compare the effects with a full term population. A controlled and randomized trial will be carried out with full term infants of adequate birth weight and preterm infants with low birth weight at 6 months of chronological or corrected age. The participants will be recruited by convenience from the charts of a Public Hospital. Participants will be randomly allocated into four groups: 1) adequate weight placebo group (AWPG); 2) adequate weight intervention group (AWIG); 2) low weight placebo group (LWPG) and 4) low weight intervention group (LWIG). . The assessor will be blinded (no knowledge of groups allocation). All infants will undergo a training program of eight sessions (2x/week; 4 weeks). The AWIG and LWIG will receive the training with an additional weight (characterized by a bracelet with a weight of 20% of the mass of the upper limbs)and the AWPG and LWPG will receive the same training, however, without the additional weight (only the bracelets).. All infants will be assessed in three different moments: 1) Pre-intervention: baseline, before the start of the intervention program; 2) Post-intervention: evaluation performed after the end of the program; and 3) Follow-up: evaluation performed seven days after the post-intervention assessment. The following kinematic dependent variables will be calculated: straightness index, mean velocity and motion units and electromyographic variables: pattern of activation and recruitment of muscle fibers - Biceps brachialis, Triceps brachialis, Deltoid and Pectoralis Major muscles; co-activation between biceps and triceps. The Qualisys Track Manager (QTM) and a wireless surface electromyography with 8-channels will be used. If normality assumptions are met, a mixed 2X2 ANOVA with repeated measures will be applied, in order to verify differences between the intervention programs, considering the dependent variables. Otherwise, non-parametric procedures of the same nature will be adopted. The significance will be set at 5% (P<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Adequate weight infants: healthy infants born with gestational age between 38-42 weeks and adequate birth weight (> 2500 grams);
* Low weight infants: healthy infants born with gestational age between 32-36 weeks and 6 days and with low birth weight (between 1500 and 2500 grams).

Exclusion Criteria:

* Anoxiated infants;
* Signs of neurological impairment (eg, hypoxic-ischemic encephalopathies grade I, II and III, intracranial hemorrhage and neonatal seizures);
* Congenital malformations (eg myelomeningocele and achondroplasias);
* Syndromes (e.g Down Syndrome);
* Sensorial alterations (visual and auditory);
* Cardiorespiratory difficulties;
* Orthopedic impairments (e.g, congenital clubfoot);
* Apgar below 8 and 10 in the first and fifth minutes, respectively.
* Infants who do not attend any of the evaluations, who do not complete at least 80% of the training or who cry uncontrollably, not allowing at least 10 reachings in the evaluations and training. Those that present intercurrences that may compromise normal neurosensorimotor development (for example, recurrent pneumonia, kidney and intestinal infection).

Ages: 6 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Movement unit | Change from Pre-Intervention (baseline) compared to Post-Intervention (4 weeks) and Follow-up (7 days)
  the number of maximum velocities between two minimum velocities, for which the difference was greater than 1 cm/s
Electromyographic activity | Change from Pre-Intervention (baseline) compared to Post-Intervention (4 weeks) and Follow-up (7 days)
  Magnitude of the muscle recruitment during the reaching behavior, measured in microvolts (root mean square - RMS)

SECONDARY OUTCOMES:
Mean Velocity | Change from Pre-Intervention (baseline) compared to Post-Intervention (4 weeks) and Follow-up (7 days)
  the ratio between the distance traveled during the reaching behavior and the duration of the movement
Straightness Index | Change from Pre-Intervention (baseline) compared to Post-Intervention (4 weeks) and Follow-up (7 days)
  ratio between the minimal distance that could have been traveled in this trajectory (distance between the initial position of the hand and the object) and the distance traveled by the hand (total trajectory). The closer is this index to 1, the straighter is the trajectory.
Grasping | Change from Pre-Intervention (baseline) compared to Post-Intervention (4 weeks) and Follow-up (7 days)
  categorical variable classified into (a) successful: when the infant was able to grasp the object with one or both hands; and (b) unsuccessful: when the infant touched the object, but did not grasp it
Muscle coactivation | Change from Pre-Intervention (baseline) compared to Post-Intervention (4 weeks) and Follow-up (7 days)
  Coactivation between the biceps and triceps muscle during the reaching behavior, measured in percentage (activation of the biceps/activation of the triceps)
Transport Unit | Change from Pre-Intervention (baseline) compared to Post-Intervention (4 weeks) and Follow-up (7 days)
  The relative duration of the first movement unit in relation to total duration of reaching
Deceleration time | Change from Pre-Intervention (baseline) compared to Post-Intervention (4 weeks) and Follow-up (7 days)
  The time necessary for the infant to decelerate the arm movement so that the hand touches an object. This period of the duration is measured from the time of appearance of the peak of velocity to the end of the reach.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Carregaro, PhD, Study Director — University of Brasilia
Locations (1):
- Campus UnB Ceilandia, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No